CLINICAL TRIAL: NCT06339619
Title: Phase II Clinical Study of Adebrelimab Combined With Apatinib and Tegafur in the Treatment of Locally Advanced or Metastatic Esophageal Squamous Cell Carcinoma That Failed First-line Immunotherapy Combined With Chemotherapy
Brief Title: Combination Immunotherapy of Adebrelimab With Apatinib and Tegafur for Immune Rechallenge Therapy in Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-1262-02
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Locally Advanced or Metastatic Esophageal Squamous Cell Carcinoma
Keywords: immunotherapy rechallenge; ESCC; Adebrelimab; Apatinib; PD-1 inhibitors; Tegafur; First-line treatment failure
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — apatinib; Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab+Apatinib+Tegafur (Experimental)
  Interventions: Drug: Adebrelimab; Drug: Apatinib; Drug: Tegafur

INTERVENTIONS:
Drug: Adebrelimab — 20mg/kg ivgtt D1 Q3W
Drug: Apatinib — 250mg PO QD
Drug: Tegafur — dosing based on body surface area：BSA<1.25m2,40mg; BSA=1.25～1.5m2,50mg; BSA>1.5m2, 60mg，PO QD D1-21 Q3W

SUMMARY:
The goal of this single-arm study is to explore the efficacy and safety of Adebrelimab in combination with Apatinib and Tegafur for the treatment of locally advanced or metastatic esophageal squamous cell carcinoma that has failed first-line standard treatment with PD-1 inhibitors in combination with chemotherapy.

DETAILED DESCRIPTION:
Background: Although immune combined chemotherapy has established its position as the first-line standard treatment for locally advanced unresectable or metastatic esophageal cancer, resistance and disease progression inevitably occur in most patients. While earlier studies have shown some therapeutic advantages of the combination of PD-1/PDL1 inhibitors with anti-angiogenic drugs, the efficacy as a second-line treatment remains unsatisfactory, necessitating further exploration of combination therapies such as chemotherapy.We conduct this single-arm study is to explore the efficacy and safety of Adebrelimab in combination with Apatinib and Tegafur in treating the patients with locally advanced or metastatic esophageal squamous cell carcinoma who has failed first-line standard treatment with PD-1 inhibitors in combination with chemotherapy.

Method: This is a prospective single arm two-stage phase II study, with an intended enrollment of 32 patients. Eligible patients with esophageal squamous cell carcinoma will receive Adebrelimab at a dose of 20mg/kg, on day 1 via intravenous drip every 21 days, in combination with Apatinib at a dose of 250mg orally once daily on days 1-21 every 21 days, and Tegafur orally once daily on days 1-21 every 21 days（BSA<1.25m2,40mg; BSA=1.25～1.5m2,50mg;BSA>1.5m2, 60mg）. Each treatment cycle lasts for 21 days. Treatment will continue until disease progression, intolerable toxicity, withdrawal of informed consent, or death. Imaging evaluation for efficacy will be conducted every 6 to 8 weeks (±7 days) after the start of the initial treatment until disease progression, death, initiation of new anticancer therapy, withdrawal of informed consent, loss to follow-up, or study termination. The primary endpoint is objective response rate (ORR), and secondary endpoints include progression-free survival (PFS), overall survival (OS), disease control rate (DCR), and safety.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old, both sexes.
2. Esophageal squamous cell carcinoma confirmed by histology or cytology with locally advanced unresectable or distant metastasis (according to AJCC 8th edition).
3. ECOG PS score of 0 ~ 1.
4. Expected survival ≥3 months.
5. Patients who have failed first-line immunotherapy combined with chemotherapy.
6. At least one measurable or unmeasurable lesion according to RECIST V1.1 criteria (subjects with intracranial lesions alone were excluded from this study).
7. Ability to swallow investigational drugs .
8. The functional level of the organ must meet the following requirements. (1) ANC≥1.5×109/L; (2) PLT≥100×109/L; (3) Hb≥90 g/L; (4) Serum albumin ≥30 g/L; (5) TBIL≤1.5×ULN; ALT and AST≤2.5 x ULN; For patients with liver metastases, ALT and AST≤5×ULN; (6) Cr ≤1.5×ULN, or creatinine clearance ≥50mL/min as calculated by the Cockcroft-Gault formula; (7) Patients with urinary protein ≥++ should undergo further 24-hour quantitative detection of urinary protein, and the detection result should be<1.0g.
9. Within 7 days prior to enrollment, women of reproductive age must confirm a negative serum pregnancy test and consent to use effective contraception during the study drug use period and within 2 months after the last dose.
10. Subjects voluntarily participate in the study after fully informed consent and sign the informed consent.

Exclusion Criteria:

1. Have been diagnosed with other malignancies within 5 years, excluding: curable carcinoma in situ of the cervix, skin basal cell carcinoma or squamous cell carcinoma, or any other tumor that has been cured .
2. Patients who had previously received treament of Adebrelimab, Apatinib or Tegafur.
3. The following conditions occurred in the previous treatment history. (1)Used Chinese medicine anti-tumor treatment within 2 weeks; (2)Received other anti-tumor therapy within 4 weeks, including but not limited to chemotherapy, radiotherapy, and targeted therapy.
4. Have not recovered from adverse events caused by prior antitumor therapy (i.e., ≤ grade 1 or at baseline).
5. Subjects who have participated in or are participating in other clinical trials within 4 weeks.
6. Received major surgery within 4 weeks or anticipated to undergo major surgery during the study period.
7. Subject is currently using a CYP3A strong inhibitor or inducer, or has discontinued a strong inhibitor for less than 5 half-lives of the medication or discontinued a strong inducer for less than 5 half-lives of the medication or 14 days (whichever is longer) before dosing.
8. Current need for treatment of central nervous system metastases or uncontrolled central nervous system metastases.
9. Risk of severe bleeding or esophageal fistula.
10. Clinically significant gastrointestinal abnormalities that may affect the intake, transport, or absorption of the drug.
11. Those with active gastrointestinal ulcers, active gastrointestinal bleeding, or perforation.
12. Within the 12 months prior to enrollment, individuals with any of the following conditions: myocardial infarction, coronary artery bypass grafting or peripheral artery bypass grafting surgery, congestive heart failure (III-IV graded by New York Heart Association), etc.; unstable angina within the 6 months prior to enrollment.
13. Within the 12 months prior to enrollment, occurrence of thrombotic events or embolic events, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, pulmonary embolism, etc., or patients currently receiving thrombolytic or anticoagulant therapy such as warfarin, heparin, or other similar medications.
14. Fridericia-corrected QT interval (QTcF)>470 ms; history of congenital long QT syndrome; history of any clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes); left ventricular ejection fraction (LVEF) <50%.
15. Those with uncontrollable pleural effusion, pericardial effusion, pelvic effusion, or ascites requiring repeated drainage.
16. Past or current interstitial lung disease or immune-related pneumonia; currently suffering from drug-induced pneumonia, radiation pneumonia requiring steroid therapy, or clinically symptomatic active pneumonia, or other moderate to severe pulmonary diseases severely affecting lung function.
17. Active infection during screening, or unexplained fever>38.5°C within 2 weeks prior to randomization.
18. Active hepatitis B or hepatitis C.
19. Received live vaccines within 4 weeks prior toenrollment and/or planned to receive live vaccines after enrollment.
20. Those with congenital or acquired immunodeficiency (such as HIV-infected individuals).
21. History of organ transplantation or allogeneic bone marrow transplantation.
22. Individuals deemed by the investigator to have other serious acute or chronic illnesses unsuitable for participation in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 6 months
  ORR is determined as the percentage of patients who had complete response (CR) or partial response (PR) as best overall response per RECIST v1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 6 months
  PFS is determined as the duration from the start of treatment until disease progression or death from any cause, whichever occurs first.
Overall survival (OS) | 12months
  OS is determined as the time from treatment to death.
≥Grade 3 AEs | 6 months
  The total incidence of grade 3 or greater adverse events was included.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China